CLINICAL TRIAL: NCT02344927
Title: A Cluster Randomised Trial of Alternative Forms of Hydration in Cancer Patients in the Last Days of Life (Feasibility Study)
Brief Title: CRT Hydration in the Last Days of Life (Feasibility Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Surrey (Other)
Collaborators: Royal Surrey County Hospital NHS Foundation Trust (Other); The Christie NHS Foundation Trust (Other); Leckhampton Hall Hospice (Cheltenham) (Unknown); Pilgrims Hospices (Kent) (Unknown); St Clare Hospice (Hastingwood) (Unknown); New Cross Hospital, Wolverhampton (Unknown); St Giles Hospice, Lichfield (Unknown); St Mary;s Hospice, Birmingham (Unknown); Velindre NHS Trust (Other Government); St Richards Hospice, Worcester (Unknown); St Catherines Hospice, Crawley (Unknown); St Margaret Hospice,Somerset (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CRC 340
Record Dates: First submitted 2014-06-04; First posted 2015-01-26 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2016-03

CONDITIONS: Cancer
Keywords: Cancer; End-of-life care; Clinically-assisted hydration
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Non-Clinically Assisted Hydration arm (Active Comparator): The interventions utilised within this trial are representative of standard clinical practice
  * Continuance of oral intake (if appropriate)
  * Regular (4 hourly) mouth care
  * Standard management of pain and other symptoms in the terminal phase.
  Interventions: Other: Non-Clinically Assisted Hydration arm
- Clinically Assisted Hydration arm (Active Comparator): The interventions utilised within this trial are representative of standard clinical practice
  * Continuance of oral intake (if appropriate)
  * Regular (4 hourly) mouth care
  * Clinically-assisted hydration
  * Standard management of pain and other symptoms in the terminal phase
  Interventions: Other: Clinically Assisted Hydration arm

INTERVENTIONS:
Other: Non-Clinically Assisted Hydration arm — Best supportive care. Continuance of oral intake (if appropriate) and regular mouth care
  Arms: Non-Clinically Assisted Hydration arm
Other: Clinically Assisted Hydration arm — Best supportive care. Continuance of oral intake (if appropriate) and regular mouth care, and clinically assisted hydration.
  Arms: Clinically Assisted Hydration arm

SUMMARY:
It is unclear whether the use of fluids given by a "drip" is beneficial to cancer patients in the last days of life, and as a result many individuals do not receive such treatment (although they do receive fluids by mouth, and regular mouth care). The researchers want to undertake a large study ("main study") to determine the benefits of fluids given by a drip, but first need to undertake a small study ("feasibility study") to ensure that the main study can be done.

The feasibility study will be done in twelve units (hospitals, hospices) in England & Wales; each unit will be allocated a treatment at random, and all patients in the unit will receive that treatment (if appropriate). Standard treatment A consists of drinking fluids (if possible), regular mouth care, and treatment of any symptoms; standard treatment B consists of drinking fluids (if possible) , regular mouth care, fluids by a drip, and treatment of any symptoms.

Patients will be assessed on a four hourly basis, and any uncontrolled symptoms will be recorded. The main symptom of interest is agitation ("delirium"), which has multiple causes, including dehydration and kidney failure. Uncontrolled symptoms will be appropriately treated, e.g. patients with pain will be given painkillers. Equally, problems relating to the fluids given by a drip will also be recorded. Involvement in the study will not interfere with the patient's general care, and there will be no additional blood or other tests.

DETAILED DESCRIPTION:
Background:

The provision of clinically-assisted hydration (CAH) at the end-of-life is one of the most contentious issues in medicine, and indeed within the general population. The reasons for contention include:

* the lack of evidence for / against CAH;
* the disparate opinions of healthcare professionals about CAH;
* the generally positive opinions of patients and their carers about CAH (and the generally negative opinions about withholding / withdrawing CAH).

It is, therefore, unsurprising that the provision of CAH at the end-of-life is extremely variable within clinical practice (i.e. 12-88% cancer patients in the last week of life).

Hypothesis:

CAH during the last days of life reduces the frequency of hyperactive delirium ("terminal agitation") in cancer patients as a result of maintenance of renal perfusion and the prevention of accumulation of toxins and drugs (i.e. prevention of dehydration).

Aims / objectives:

The aim of the definitive study is to evaluate the utility / role of CAH in cancer patients in the last days of life.

The aim of the feasibility study is to answer the question "can this study (the definitive study) be done".

The objectives of the feasibility study are to:

* assess the recruitment rate, i.e. number eligible patients, number recruited patients, barriers to recruitment;
* assess the retention rate;
* assess impact of trial procedures on clinical workload, i.e. completion of clinical assessment documentation, undertaking mouth care / CAH;
* assess the adequacy of resources to conduct the study at research centres;
* assess the adequacy of resources to support the study at Surrey Clinical Research Centre;
* determine other challenges for researchers / research centres;
* determine other challenges for Surrey Clinical Research Centre;
* assess safety of CAH
* determine total variability / intra-cluster correlation coefficient

Methodology:

The study is a cluster randomised trial with a mixed method of consenting. Consent sought from patients (whenever possible), or advice from a "personal consultee" (when a patient is unable to provide consent), or from a "nominated consultee" (when a patient is unable to provide consent, and there is no personal consultee).

Sites will be randomised to either "standard intervention arm A", or "standard intervention arm B". Patients in standard intervention arm A will be managed with continuance of oral intake (if appropriate), and regular "mouth care". Mouth care will be performed at least every four hours, and will correspond to the investigational site's policy / procedures for oral care in the terminal phase. Patients in standard intervention arm B will be managed with continuance of oral intake (if appropriate), regular "mouth care", and CAH, i.e. parenteral fluids. Again, mouth care will be performed at least every four hours, and will correspond to the investigational site's policy / procedures for oral care in the terminal phase. The parenteral fluids may be administered either intravenously or subcutaneously at the discretion of the medical and nursing team. The type of fluid to be administered will be dextrose saline (i.e. 4% dextrose, 0.18% sodium chloride), and the volume to be administered will be dependent on the patient's weight.

The primary endpoint of the definitive study is the frequency of hyperactive delirium ("terminal agitation"), and this will be assessed using the Modified Richmond Agitation and Sedation Scale (administered every four hours). Other data to be collected include the frequency of pain, respiratory secretions / "death rattle", dyspnoea, nausea and vomiting, adverse effects from the CAH, and overall survival. In addition, data will be collected on the use of anti-psychotic drugs, sedative drugs, analgesics, anti-secretory drugs, and other end-of-life medication.

A "cluster representation mechanism" (CRM) will be utilised, including the appointment of site-specific "study guardians" and "study gatekeepers", who will protect and respect the rights of the cluster and the individual participants within the cluster.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of cancer
* Age ≥ 18 yr
* Estimated prognosis of ≤ 1 week
* Patient unable to maintain sufficient oral intake (1L / day)

Exclusion criteria:

* Patient clinically dehydrated
* Patient has hyperactive delirium ("terminal agitation") at present
* Patient has had hyperactive delirium ("terminal agitation") in the last 24hr
* Clinical indication for clinically-assisted hydration (e.g. hypercalcaemia)
* Clinical contra-indication to clinically-assisted hydration (e.g. cardiac failure)
* Clinical contra-indication to peripheral cannulation
* Intravenous fluids / subcutaneous fluids / total parenteral nutrition (TPN) / enteral feeding or fluids already being administered
* Patient likely to be transferred to another setting for end of life care (e.g. home, hospice)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2015-02; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | Up to 12 months
  Sample size is 200

SECONDARY OUTCOMES:
Retention (% participants complete the study in a one year period) | Up to 12 months
  > 67% participants complete the study in a one year period
Adherence (% nursing observation completed in a one year period) | Up to 12 months
  >67% nursing observation completed in a one year period
Treatment related adverse events | Up to 12 months
  <50% participants have clinically assisted hydration discontinued due to treatment- related adverse events, in a one year period

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Davies, Principal Investigator — Royal Surrey County Hospital NHS Foundation Trust
Locations (12):
- United Kingdom (12):
  - St Clare Hospice, Harlow, Essex
  - Leckampton Hall Hospice, Cheltenham, Gloucestershire
  - Pilgrims Hospice, Canterbury, Kent
  - The Christie NHS Foundation Trust, Manchester, Lancashire
  - New Cross Hospital, Wolverhampton, Midlands
  - St Margaret's Hospice, Taunton, Somerset
  - St Giles Hospice, Lichfield, Staffordshire
  - The Royal Surrey County Hospital NHS Foundation Trust, Guildford, Surrey
  - St Catherine's Hospice, Crawley, Sussex
  - St Mary Hospice, Birmingham, West Midlands
  - St Richards Hospice, Worcester, Worcestershire
  - Velindre Cancer centre, Cardiff

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Davies AN, Waghorn M, Webber K, Johnsen S, Mendis J, Boyle J. A cluster randomised feasibility trial of clinically assisted hydration in cancer patients in the last days of life. Palliat Med. 2018 Apr;32(4):733-743. doi: 10.1177/0269216317741572. Epub 2018 Jan 18. PMID 29343167
- [Derived] Davies A, Waghorn M, Boyle J, Gallagher A, Johnsen S. Alternative forms of hydration in patients with cancer in the last days of life: study protocol for a randomised controlled trial. Trials. 2015 Oct 14;16:464. doi: 10.1186/s13063-015-0988-3. PMID 26466809